CLINICAL TRIAL: NCT01531413
Title: Single-Blind, Randomized, Controlled Trial of Oxygen Insufflation to Reduce Incidence of Postoperative Abscess in Laparoscopic Appendectomy
Brief Title: Oxygen Insufflation To Reduce Postoperative Abscess In Laparoscopic Appendectomy
Acronym: AppyO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang, Steve S., M.D. (Individual)
Collaborators: Santa Barbara Cottage Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: AppyO2_SBCH
Record Dates: First submitted 2012-02-07; First posted 2012-02-13 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Postoperative Abscess
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxygen Insufflation (Experimental): At the end of the laparoscopic appendectomy we will desufflate the abdomen of CO2 then reinsufflate with oxygen to washout the CO2 leaving an oxygen rich environment
  Interventions: Other: Oxygen Insufflation

INTERVENTIONS:
Other: Oxygen Insufflation — At the end of the case, abdomen will be desufflated with CO2 then insufflated with oxygen
  Other Names: Oxygen

SUMMARY:
Oxygen has inherent bactericidal properties. The investigators are testing to see if they can reduce the incidence of postoperative abscesses following laparoscopic appendectomy by insufflating with oxygen at the end of the case.

DETAILED DESCRIPTION:
Intra-abdominal abscess a well-known complication of both open and laparoscopic appendectomy, especially in the setting of perforated and gangrenous appendicitis. The reviewed literature cites an incidence of about 10%. Besides peri-operative antibiotic administration there have been few developments to reduce this inherent risk. Oxygen rich environments are potently bactericidal, and thus it is our hypothesis that establishing an oxygen rich ambience within the abdomen at the conclusion of laparoscopy could curtail bacterial growth and subsequent abscess formation.

In the experimental arm, at the conclusion of all surgical dissection and manipulation, the carbon dioxide insufflate will be exchanged with oxygen to generate a high intra-abdominal concentration. Oxygen will be infused for 15 seconds as CO2 is allowed to escape through the open trocars. In the control arm Co2 will be allowed to escape through the open trocar ports without any oxygen flush. Patients will receive a standardized operation as well as standard post-operative care and follow up.

ELIGIBILITY:
Inclusion Criteria:

* Nonpregnant adults 18 or older
* Clinical or image proven appendicitis
* Undergoing Laparoscopic Appendectomy

Exclusion Criteria:

* Any pregnant females
* Anyone under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Postoperative Abscess | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steve S Chang, MD, Principal Investigator — Santa Barbara Cottage Hospital
Locations (1):
- Santa Barbara Cottage Hospital, Santa Barbara, California, United States